CLINICAL TRIAL: NCT03096444
Title: Antipruritic Effect of Topical Ketamine, Amitriptyline, and Lidocaine
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Efficacy was not seen after interim analysis
Sponsor: Gil Yosipovitch (Other)
Responsible Party: Sponsor-Investigator, Gil Yosipovitch, Professor, University of Miami
Organization: University of Miami (Other)
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: 20170087
Record Dates: First submitted 2017-03-16; First posted 2017-03-30 (Actual); Results first posted 2019-07-02 (Actual); Last update posted 2019-07-02 (Actual); Status verified 2019-04

CONDITIONS: Pruritus
MeSH Terms: conditions — Pruritus | interventions — Ketamine; Amitriptyline; Lidocaine

STUDY DESIGN:
Intervention Model Description: The antipruritic effect of 4 topical treatments and 1 vehicle treatment will be explored in each subject. Study visit 1 will consist of testing 3 topical formulations, and study visit 2 will test the remaining 2 topical formulations in each subject.
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (5):
- Topical KeAmLi combo (Experimental): Topical KeAmLi-combo (ketamine 10%, amitriptyline 5%, and lidocaine 5%) will be applied to one four 4 x 4 cm predefined skin areas on the ventral forearms during one of two study visits. The pre-treatment will occur under topical occlusion for 30 minutes to allow the ointment to be adsorbed. Following this, residual ointment will be removed and sensory testing, strictly within the pretreated area, will commence.
  Interventions: Combination Product: Ketamine hydrochloride, Amitriptyline hydrochloride, and Lidocaine hydrochloride
- Topical ketamine (Experimental): Topical ketamine 10% will be applied to one four 4 x 4 cm predefined skin areas on the ventral forearms during one of two study visits. The pre-treatment will occur under topical occlusion for 30 minutes to allow the ointment to be adsorbed. Following this, residual ointment will be removed and sensory testing, strictly within the pretreated area, will commence.
  Interventions: Drug: Ketamine Hydrochloride
- Topical amitriptyline (Experimental): Topical amitriptyline 5% will be applied to one four 4 x 4 cm predefined skin areas on the ventral forearms during one of two study visits. The pre-treatment will occur under topical occlusion for 30 minutes to allow the ointment to be adsorbed. Following this, residual ointment will be removed and sensory testing, strictly within the pretreated area, will commence.
  Interventions: Drug: Amitriptyline Hydrochloride
- Topical lidocaine (Experimental): Topical lidocaine 5% will be applied to one four 4 x 4 cm predefined skin areas on the ventral forearms during one of two study visits. The pre-treatment will occur under topical occlusion for 30 minutes to allow the ointment to be adsorbed. Following this, residual ointment will be removed and sensory testing, strictly within the pretreated area, will commence.
  Interventions: Drug: Lidocaine Hydrochloride
- Topical vehicle (Placebo Comparator): Topical vehicle (PCCA Lipoderm) will be applied to one four 4 x 4 cm predefined skin areas on the ventral forearms during one of two study visits. The pre-treatment will occur under topical occlusion for 30 minutes to allow the ointment to be adsorbed. Following this, residual ointment will be removed and sensory testing, strictly within the pretreated area, will commence.
  Interventions: Drug: Lipoderm Cream

INTERVENTIONS:
Drug: Ketamine Hydrochloride — 2g of topical 10% Ketamine will be applied for 30 minutes on one 4x4cm area on the volar forearm in one of two study visits.
  Other Names: Topical ketamine
  Arms: Topical ketamine
Drug: Amitriptyline Hydrochloride — 2g of topical 5% Amitriptyline will be applied for 30 minutes on one 4x4cm area on the volar forearm in one of two study visits.
  Other Names: Topical amitriptyline
  Arms: Topical amitriptyline
Drug: Lidocaine Hydrochloride — 2g of topical 5% Lidocaine will be applied for 30 minutes on one 4x4cm area on the volar forearm in one of two study visits.
  Other Names: Topical lidocaine
  Arms: Topical lidocaine
Combination Product: Ketamine hydrochloride, Amitriptyline hydrochloride, and Lidocaine hydrochloride — 2g of topical KeAmLi-combo (ketamine 10%, amitriptyline 5%, and lidocaine 5%) will be applied for 30 minutes on one 4x4cm area on the volar forearm in one of two study visits.
  Other Names: Topical KeAmLi combo
  Arms: Topical KeAmLi combo
Drug: Lipoderm Cream — 2g of topical vehicle (Lipoderm) will be applied for 30 minutes on one 4x4cm area on the volar forearm in one of two study visits.
  Other Names: Topical vehicle
  Arms: Topical vehicle

SUMMARY:
The purpose of this study is to examine the antipruritic efficacy of topical ketamine, amitriptyline, lidocaine, and a tri-combination of ketamine, amitriptyline and lidocaine (hereafter referred to as "KeAmLi") using non-histaminergic itch provocations in healthy volunteers. The primary outcome is itch reduction (AUC) between the vehicle and active treatment (KeAmLi-combo). Secondary outcomes include modality-specific analgesic properties of the topically applied ketamine, amitriptyline, lidocaine, and KeAmLi-combo to controlled quantitative thermal and mechanical stimuli, which can improve our understanding of the mechanism of action of these substances in the context of topical therapy.

DETAILED DESCRIPTION:
This is a double-blind, vehicle-controlled study to evaluate the antipruritic efficacy of topical ketamine, amitriptyline, lidocaine, and a tri-combination of ketamine, amitriptyline and lidocaine (hereafter referred to as "KeAmLi") using non-histaminergic itch provocations in healthy volunteers. Each participant will be pre-treated with the vehicle and 4 active topical creams, over two study visits (3 treatments on the 1st visit and 2 treatment on the 2nd visit). Each treatment will be applied to the randomized forearm test area for 30 minute, and then sensory testing will be performed. Sensory testing includes thermal and mechanical stimuli, and itch induction using the plant cowhage. These tests will reveal mechanistic information and potential cellular and molecular targets for improved antipruritic and analgesic therapies.

ELIGIBILITY:
Inclusion Criteria:

1. Healthy subjects (absence of disease) between 18 and 50 years of age.
2. Must be in general good health with no disease or physical conditions that would impair evaluation of itch and pain perception.
3. No history of chronic itch or pain.
4. Must abstain from the use of any systemic or topical anti-histamine, steroid, or pain relief medications 48 hours prior to the study visits.
5. Must abstain from the use of moisturizers on the arms the day of study visit.

Exclusion Criteria:

1. Individuals under 18 or over 50 years of age.
2. Inability to complete the required measures.
3. The presence of an itchy skin disease or a painful condition.
4. Diagnosis of diseased that would affect itch or pain perception (e.g. neuropathies).
5. Currently enrolled in any investigational study in which the subject is receiving any type of drug, biological, or non-drug therapy.
6. Use of oral, topical analgesics, or other medications known to interfere with itch or pain perception 48 hours prior to the study visits (e.g. antihistamines, anesthetics, anti-inflammatories, opioids, neuroleptics, etc.).
7. Use of emollients on the volar aspects of the forearms arms on the day of the study visit.
8. Use of anti-depressants, anti-psychotics, and illicit drugs.
9. Known history of neuropathy, uremia, uncontrolled thyroid disease, and diabetes mellitus.
10. Known history of anaphylactic shock, or allergy to cowhage and/or known adverse reactions to lidocaine (or other local anesthetics of the amide type), ketamine or amitriptyline.

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 13 (Actual)
Dates: Start 2017-05-23 (Actual); Primary Completion 2017-07-19 (Actual); Study Completion 2017-07-21 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Gil Yosipovitch, MD, Principal Investigator — University of Miami
Locations (1):
- University of Miami, Miami, Florida, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Weisshaar E, Gieler U, Kupfer J, Furue M, Saeki H, Yosipovitch G; International Forum on the Study of Itch. Questionnaires to assess chronic itch: a consensus paper of the special interest group of the International Forum on the Study of Itch. Acta Derm Venereol. 2012 Sep;92(5):493-6. doi: 10.2340/00015555-1402. PMID 22688895
- [Background] Matterne U, Apfelbacher CJ, Vogelgsang L, Loerbroks A, Weisshaar E. Incidence and determinants of chronic pruritus: a population-based cohort study. Acta Derm Venereol. 2013 Sep 4;93(5):532-7. doi: 10.2340/00015555-1572. PMID 23450324
- [Background] Matterne U, Apfelbacher CJ, Loerbroks A, Schwarzer T, Buttner M, Ofenloch R, Diepgen TL, Weisshaar E. Prevalence, correlates and characteristics of chronic pruritus: a population-based cross-sectional study. Acta Derm Venereol. 2011 Oct;91(6):674-9. doi: 10.2340/00015555-1159. PMID 21879245
- [Background] Leknes SG, Bantick S, Willis CM, Wilkinson JD, Wise RG, Tracey I. Itch and motivation to scratch: an investigation of the central and peripheral correlates of allergen- and histamine-induced itch in humans. J Neurophysiol. 2007 Jan;97(1):415-22. doi: 10.1152/jn.00070.2006. Epub 2006 Aug 16. PMID 16914620
- [Background] Wahlgren CF. Itch and atopic dermatitis: an overview. J Dermatol. 1999 Nov;26(11):770-9. doi: 10.1111/j.1346-8138.1999.tb02090.x. PMID 10635621
- [Background] Brenaut E, Garlantezec R, Talour K, Misery L. Itch characteristics in five dermatoses: non-atopic eczema, atopic dermatitis, urticaria, psoriasis and scabies. Acta Derm Venereol. 2013 Sep 4;93(5):573-4. doi: 10.2340/00015555-1599. No abstract available. PMID 23722181
- [Background] Carroll CL, Balkrishnan R, Feldman SR, Fleischer AB Jr, Manuel JC. The burden of atopic dermatitis: impact on the patient, family, and society. Pediatr Dermatol. 2005 May-Jun;22(3):192-9. doi: 10.1111/j.1525-1470.2005.22303.x. PMID 15916563
- [Background] Patel T, Yosipovitch G. Therapy of pruritus. Expert Opin Pharmacother. 2010 Jul;11(10):1673-82. doi: 10.1517/14656566.2010.484420. PMID 20426711
- [Background] Kopsky DJ, Keppel Hesselink JM, Bhaskar A, Hariton G, Romanenko V, Casale R. Analgesic effects of topical ketamine. Minerva Anestesiol. 2015 Apr;81(4):440-9. Epub 2014 May 22. PMID 24847738
- [Background] Coggeshall RE, Carlton SM. Ultrastructural analysis of NMDA, AMPA, and kainate receptors on unmyelinated and myelinated axons in the periphery. J Comp Neurol. 1998 Feb 2;391(1):78-86. doi: 10.1002/(sici)1096-9861(19980202)391:13.3.co;2-8. PMID 9527543
- [Background] Carlton SM, Coggeshall RE. Inflammation-induced changes in peripheral glutamate receptor populations. Brain Res. 1999 Feb 27;820(1-2):63-70. doi: 10.1016/s0006-8993(98)01328-6. PMID 10023031
- [Background] Davidson EM, Coggeshall RE, Carlton SM. Peripheral NMDA and non-NMDA glutamate receptors contribute to nociceptive behaviors in the rat formalin test. Neuroreport. 1997 Mar 3;8(4):941-6. doi: 10.1097/00001756-199703030-00025. PMID 9141069
- [Background] Mehta AK, Halder S, Khanna N, Tandon OP, Singh UR, Sharma KK. Role of NMDA and opioid receptors in neuropathic pain induced by chronic constriction injury of sciatic nerve in rats. J Basic Clin Physiol Pharmacol. 2012;23(2):49-55. doi: 10.1515/jbcpp-2012-0003. PMID 23091273
- [Background] Zhou S, Bonasera L, Carlton SM. Peripheral administration of NMDA, AMPA or KA results in pain behaviors in rats. Neuroreport. 1996 Mar 22;7(4):895-900. doi: 10.1097/00001756-199603220-00012. PMID 8724668
- [Background] Tandon OP, Mehta AK, Halder S, Khanna N, Sharma KK. Peripheral interaction of opioid and NMDA receptors in inflammatory pain in rats. Indian J Physiol Pharmacol. 2010 Jan-Mar;54(1):21-31. PMID 21046916
- [Background] Sandroni P, Davis MD. Combination gel of 1% amitriptyline and 0.5% ketamine to treat refractory erythromelalgia pain: a new treatment option? Arch Dermatol. 2006 Mar;142(3):283-6. doi: 10.1001/archderm.142.3.283. No abstract available. PMID 16549702
- [Background] Gerner P, Kao G, Srinivasa V, Narang S, Wang GK. Topical amitriptyline in healthy volunteers. Reg Anesth Pain Med. 2003 Jul-Aug;28(4):289-93. doi: 10.1016/s1098-7339(03)00209-8. PMID 12945021
- [Background] Lynch ME, Clark AJ, Sawynok J, Sullivan MJ. Topical amitriptyline and ketamine in neuropathic pain syndromes: an open-label study. J Pain. 2005 Oct;6(10):644-9. doi: 10.1016/j.jpain.2005.04.008. PMID 16202956
- [Background] Uzaraga I, Gerbis B, Holwerda E, Gillis D, Wai E. Topical amitriptyline, ketamine, and lidocaine in neuropathic pain caused by radiation skin reaction: a pilot study. Support Care Cancer. 2012 Jul;20(7):1515-24. doi: 10.1007/s00520-011-1240-7. Epub 2011 Aug 17. PMID 21847539
- [Background] Griffin JR, Davis MD. Amitriptyline/Ketamine as therapy for neuropathic pruritus and pain secondary to herpes zoster. J Drugs Dermatol. 2015 Feb;14(2):115-8. PMID 25689805
- [Background] Lynch ME, Clark AJ, Sawynok J. A pilot study examining topical amitriptyline, ketamine, and a combination of both in the treatment of neuropathic pain. Clin J Pain. 2003 Sep-Oct;19(5):323-8. doi: 10.1097/00002508-200309000-00007. PMID 12966259
- [Background] LaMotte RH, Dong X, Ringkamp M. Sensory neurons and circuits mediating itch. Nat Rev Neurosci. 2014 Jan;15(1):19-31. doi: 10.1038/nrn3641. PMID 24356071
- [Background] Sawynok J. Topical analgesics for neuropathic pain in the elderly: current and future prospects. Drugs Aging. 2014 Dec;31(12):853-62. doi: 10.1007/s40266-014-0218-9. PMID 25373920
- [Background] Schmelz M, Schmidt R, Bickel A, Handwerker HO, Torebjork HE. Specific C-receptors for itch in human skin. J Neurosci. 1997 Oct 15;17(20):8003-8. doi: 10.1523/JNEUROSCI.17-20-08003.1997. PMID 9315918
- [Background] Abels C. Intra-epidermal nerve fibres in human skin: back to the roots. Exp Dermatol. 2014 Apr;23(4):232-3. doi: 10.1111/exd.12326. Epub 2014 Feb 16. PMID 24450967
- [Background] Zylka MJ, Rice FL, Anderson DJ. Topographically distinct epidermal nociceptive circuits revealed by axonal tracers targeted to Mrgprd. Neuron. 2005 Jan 6;45(1):17-25. doi: 10.1016/j.neuron.2004.12.015. PMID 15629699
- [Background] Namer B, Carr R, Johanek LM, Schmelz M, Handwerker HO, Ringkamp M. Separate peripheral pathways for pruritus in man. J Neurophysiol. 2008 Oct;100(4):2062-9. doi: 10.1152/jn.90482.2008. Epub 2008 Jun 18. PMID 18562548
- [Background] Stander S, Schmelz M. Chronic itch and pain--similarities and differences. Eur J Pain. 2006 Jul;10(5):473-8. doi: 10.1016/j.ejpain.2006.03.005. Epub 2006 May 5. PMID 16678456
- [Background] Lynch ME, Clark AJ, Sawynok J, Sullivan MJ. Topical 2% amitriptyline and 1% ketamine in neuropathic pain syndromes: a randomized, double-blind, placebo-controlled trial. Anesthesiology. 2005 Jul;103(1):140-6. doi: 10.1097/00000542-200507000-00021. PMID 15983466
- [Background] Tey HL, Yosipovitch G. Targeted treatment of pruritus: a look into the future. Br J Dermatol. 2011 Jul;165(1):5-17. doi: 10.1111/j.1365-2133.2011.10217.x. Epub 2011 May 30. PMID 21219293
- [Background] Hoeck EA, Marker JB, Gazerani P, H Andersen H, Arendt-Nielsen L. Preclinical and human surrogate models of itch. Exp Dermatol. 2016 Oct;25(10):750-7. doi: 10.1111/exd.13078. PMID 27194117
- [Background] Andersen HH, Sorensen AR, Nielsen GA, Molgaard MS, Stilling P, Boudreau SA, Elberling J, Arendt-Nielsen L. A Test-Retest Reliability Study of Human Experimental Models of Histaminergic and Non-histaminergic Itch. Acta Derm Venereol. 2017 Feb 8;97(2):198-207. doi: 10.2340/00015555-2502. PMID 27377123
- [Background] Rolke R, Baron R, Maier C, Tolle TR, Treede -DR, Beyer A, Binder A, Birbaumer N, Birklein F, Botefur IC, Braune S, Flor H, Huge V, Klug R, Landwehrmeyer GB, Magerl W, Maihofner C, Rolko C, Schaub C, Scherens A, Sprenger T, Valet M, Wasserka B. Quantitative sensory testing in the German Research Network on Neuropathic Pain (DFNS): standardized protocol and reference values. Pain. 2006 Aug;123(3):231-243. doi: 10.1016/j.pain.2006.01.041. Epub 2006 May 11. PMID 16697110
- [Background] Sikand P, Shimada SG, Green BG, LaMotte RH. Similar itch and nociceptive sensations evoked by punctate cutaneous application of capsaicin, histamine and cowhage. Pain. 2009 Jul;144(1-2):66-75. doi: 10.1016/j.pain.2009.03.001. Epub 2009 May 6. PMID 19423224
- [Background] LaMotte RH, Shimada SG, Green BG, Zelterman D. Pruritic and nociceptive sensations and dysesthesias from a spicule of cowhage. J Neurophysiol. 2009 Mar;101(3):1430-43. doi: 10.1152/jn.91268.2008. Epub 2009 Jan 14. PMID 19144738
- [Background] Sikand P, Shimada SG, Green BG, LaMotte RH. Sensory responses to injection and punctate application of capsaicin and histamine to the skin. Pain. 2011 Nov;152(11):2485-2494. doi: 10.1016/j.pain.2011.06.001. Epub 2011 Jul 29. PMID 21802851
- [Background] Papoiu AD, Coghill RC, Kraft RA, Wang H, Yosipovitch G. A tale of two itches. Common features and notable differences in brain activation evoked by cowhage and histamine induced itch. Neuroimage. 2012 Feb 15;59(4):3611-23. doi: 10.1016/j.neuroimage.2011.10.099. Epub 2011 Nov 12. PMID 22100770
- [Background] Rolke R, Magerl W, Campbell KA, Schalber C, Caspari S, Birklein F, Treede RD. Quantitative sensory testing: a comprehensive protocol for clinical trials. Eur J Pain. 2006 Jan;10(1):77-88. doi: 10.1016/j.ejpain.2005.02.003. PMID 16291301
- [Background] Reddy VB, Iuga AO, Shimada SG, LaMotte RH, Lerner EA. Cowhage-evoked itch is mediated by a novel cysteine protease: a ligand of protease-activated receptors. J Neurosci. 2008 Apr 23;28(17):4331-5. doi: 10.1523/JNEUROSCI.0716-08.2008. PMID 18434511
- [Background] Maier C, Baron R, Tolle TR, Binder A, Birbaumer N, Birklein F, Gierthmuhlen J, Flor H, Geber C, Huge V, Krumova EK, Landwehrmeyer GB, Magerl W, Maihofner C, Richter H, Rolke R, Scherens A, Schwarz A, Sommer C, Tronnier V, Uceyler N, Valet M, Wasner G, Treede DR. Quantitative sensory testing in the German Research Network on Neuropathic Pain (DFNS): somatosensory abnormalities in 1236 patients with different neuropathic pain syndromes. Pain. 2010 Sep;150(3):439-450. doi: 10.1016/j.pain.2010.05.002. PMID 20627413
- [Background] Mainka T, Malewicz NM, Baron R, Enax-Krumova EK, Treede RD, Maier C. Presence of hyperalgesia predicts analgesic efficacy of topically applied capsaicin 8% in patients with peripheral neuropathic pain. Eur J Pain. 2016 Jan;20(1):116-29. doi: 10.1002/ejp.703. Epub 2015 Apr 8. PMID 25854794
- [Background] Tam E, Furlan AD. Transdermal lidocaine and ketamine for neuropathic pain: a study of effectiveness and tolerability. Open Neurol J. 2012;6:58-64. doi: 10.2174/1874205X01206010058. Epub 2012 Jun 28. PMID 22833771
- [Background] Gammaitoni A, Gallagher RM, Welz-Bosna M. Topical ketamine gel: possible role in treating neuropathic pain. Pain Med. 2000 Mar;1(1):97-100. doi: 10.1046/j.1526-4637.2000.00006.x. PMID 15101968
- [Background] Sullivan RW, Ryzewski M, Holland MG, Marraffa JM. Compounded ointment results in severe toxicity in a pediatric patient. Pediatr Emerg Care. 2013 Nov;29(11):1220-2. doi: 10.1097/PEC.0b013e3182aa4748. PMID 24196095
- [Background] Jackson D, Chen AH, Bennett CR. Identifying true lidocaine allergy. J Am Dent Assoc. 1994 Oct;125(10):1362-6. doi: 10.14219/jada.archive.1994.0180. PMID 7844301
- [Background] Taddio A, Ohlsson A, Einarson TR, Stevens B, Koren G. A systematic review of lidocaine-prilocaine cream (EMLA) in the treatment of acute pain in neonates. Pediatrics. 1998 Feb;101(2):E1. doi: 10.1542/peds.101.2.e1. PMID 9445511
- [Background] Gammaitoni AR, Alvarez NA, Galer BS. Safety and tolerability of the lidocaine patch 5%, a targeted peripheral analgesic: a review of the literature. J Clin Pharmacol. 2003 Feb;43(2):111-7. doi: 10.1177/0091270002239817. PMID 12616661
- [Background] Selcuk E, Erturk S, Afrashi A. An adverse reaction to local anaesthesia: report of a case. Dent Update. 1996 Oct;23(8):345-6. PMID 9452627
- [Background] Friedman PM, Mafong EA, Friedman ES, Geronemus RG. Topical anesthetics update: EMLA and beyond. Dermatol Surg. 2001 Dec;27(12):1019-26. doi: 10.1046/j.1524-4725.2001.01855.x. PMID 11849263
- [Background] Papoiu AD, Tey HL, Coghill RC, Wang H, Yosipovitch G. Cowhage-induced itch as an experimental model for pruritus. A comparative study with histamine-induced itch. PLoS One. 2011 Mar 14;6(3):e17786. doi: 10.1371/journal.pone.0017786. PMID 21423808

RESULTS

PARTICIPANT FLOW:
Units Other Than Participants: 4x4cm skin arm test area
Groups:
- Topical KeAmLi Combo/Ketamine/Amitriptyline/Lidocaine/Vehicle: Each participant will receive topical cream treatments applied for 30 minutes to 5 separate 4 x 4 cm predefined skin areas on the ventral forearms.
  The 5 topical treatments are:
  Topical KeAmLi Combo: Ketamine hydrochloride, Amitriptyline hydrochloride, and Lidocaine hydrochloride: 2g of topical KeAmLi-combo (ketamine 10%, amitriptyline 5%, and lidocaine 5%) Topical ketamine: 10% Topical amitriptyline: 5% Topical lidocaine: 5% Topical vehicle: PCCA Lipoderm cream
Period: Overall Study
Arm/Group | Topical KeAmLi Combo/Ketamine/Amitriptyline/Lidocaine/Vehicle
Started | 13; 65 4x4cm skin arm test area
Completed | 13; 65 4x4cm skin arm test area
Not Completed | 0; 0 4x4cm skin arm test area

BASELINE CHARACTERISTICS:
Population: All subjects received 5 topical cream treatments
Units Other Than Participants: arm skin test area
Arm/Group | Topical KeAmLi Combo/Ketamine/Amitriptyline/Lidocaine/Vehicle
Number analyzed (Participants) | 13
Number analyzed (arm skin test area) | 65
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 13
  >=65 years | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 9
  Male | 4
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 5
  Not Hispanic or Latino | 8
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 3
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 1
  White | 9
  More than one race | 0
  Unknown or Not Reported | 0

OUTCOME MEASURES:

1. Primary Outcome: Peak Itch Intensity Between the Vehicle and Active Treatments (Individual and KeAmLi-combo).
Description: Peak itch intensity between the vehicle and 4 other active treatments (individual ketamine, amitriptyline, or lidocaine, and KeAmLi-combo). Itch intensity was measured on a 100mm scale visual analog scale for 10 minutes. 0 was weighted with "no itch" and 100 was weighted with "most itch imaginable".
Time Frame: 10 minutes
Population: All subjects received 5 topical cream treatments.
Measure: Mean (Standard Deviation); unit: Intensity score
Arm/Group | Topical KeAmLi Combo | Topical Ketamine | Topical Amitriptyline | Topical Lidocaine | Topical Vehicle
Number analyzed (Participants) | 13 | 13 | 13 | 13 | 13
Intensity score | 62.7 (29.00397851) | 63.1 (30.11218341) | 69.2 (29.52725816) | 65.8 (33.80866222) | 61.9 (33.95207784)

2. Secondary Outcome: Thermal Threshold Detection (Warmth and Heat Pain)
Description: Two standardized quantitative sensory tests are performed to measure warmth detection threshold (assesses the threshold of which warmth sensation is first detected) and heat pain threshold (assesses the threshold at which heat pain sensation is first detected). Measured in change in celsius.
Time Frame: 3 minutes
Population: All subjects received treatment with the 5 topical cream formulations. Quantitative sensory testing was performed on each area of treated skin.
Measure: Mean (Standard Deviation); unit: Degrees celsius
Arm/Group | Topical KeAmLi Combo | Topical Ketamine | Topical Amitriptyline | Topical Lidocaine | Topical Vehicle
Number analyzed (Participants) | 13 | 13 | 13 | 13 | 13
Degrees celsius
  Warm Detection Threshold | 33.6 (0.303939003) | 34.0 (1.10853976) | 33.9 (0.649150223) | 33.7 (0.389004867) | 33.8 (0.577436619)
  Heat Pain Threshold | 39.8 (2.401845207) | 40.0 (2.2098072) | 40.0 (2.80388162) | 39.4 (2.305045253) | 39.7 (2.227588606)

3. Secondary Outcome: Mechanical Thresholds (Mechanical Detection and Pain).
Description: Assess mechanical detection and pain thresholds using von Frey filaments stimulators (measured in force mN) to calculate the final threshold as the geometric mean of five series of ascending and descending stimuli.
Time Frame: 5 minutes
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: mN
Arm/Group | Topical KeAmLi Combo | Topical Ketamine | Topical Amitriptyline | Topical Lidocaine | Topical Vehicle
Number analyzed (Participants) | 13 | 13 | 13 | 13 | 13
mN
  Mechanical Detection Threshold | 3.519376956 (0.122225324) | 3.464204768 (0.16205246) | 3.573423965 (0.141531726) | 3.546037659 (0.157416303) | 3.525692637 (0.169487169)
  Mechanical Pain Threshold | 152.3293608 (90.32609423) | 135.9 (121.5234567) | 152.4768146 (114.1149716) | 126.9 (106.9414678) | 148.7138273 (104.3418768)

ADVERSE EVENTS:
Time Frame: Data was collect for 1 week from the time of treatment.
Arm/Group | Topical KeAmLi Combo | Topical Ketamine | Topical Amitriptyline | Topical Lidocaine | Topical Vehicle
All-Cause Mortality (participants affected / at risk) | 0/13 | 0/13 | 0/13 | 0/13 | 0/13
Serious Adverse Events (participants affected / at risk) | 0/13 | 0/13 | 0/13 | 0/13 | 0/13
Other Adverse Events (participants affected / at risk) | 0/13 | 0/13 | 0/13 | 0/13 | 0/13

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2017-03-29): https://cdn.clinicaltrials.gov/large-docs/44/NCT03096444/Prot_SAP_000.pdf